CLINICAL TRIAL: NCT03558776
Title: Influence of the Background Diet on Metabolism of Land-based n-3 PUFA From Linseed Oil - Focus: Conversion of Alpha Linolenic Acid (ALA; KoALA Study)
Brief Title: Influence of the Background Diet on Metabolism of Land-based n-3 PUFA
Acronym: KoALA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Christine Dawczynski,PhD, Leader of the Junior Research Group Nutritional Concepts, University of Jena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H6_18
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2018-06

CONDITIONS: Endogenous Conversion of Alpha Linolenic Acid
Keywords: alpha linolenic acid, linseed oil, eicosapentaenoic acid, docosahexaenoic acid
MeSH Terms: interventions — Linseed Oil

STUDY DESIGN:
Intervention Model Description: Blood samples will be taken at the beginning and regularly every four weeks during the 12-weeks intervention period. For all groups, the consumption of additional n-3 PUFA sources is not permitted during the entire intervention period. The study intervention will consist of a daily dose of linseed oil (LO, 10 En%) and prepared daily menu plans determining the background diet, except for the control group D. The fat composition of the developed daily menu plans (fat content 20 En%) will differ between the groups A to C. For groups A to C, the daily menu plans will ensure an adequate intake of energy and nutrients according to the guidelines of the German Society of Nutrition. Group D serves as control because in this group the background diet is not fixed by menu plans. Participants of group D must follow their normal dietary habits, i.e. a typical Western diet (LA intake is about 15 g/d (5-7 En%) / SFA intake ranges from 10 to 15 En%).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Linseed oil plus defined background diet (high linolec acid) (Active Comparator): Linseed oil (LO) plus daily menu plans (total dietary fat intake: 30 En%): 10 En% LO plus menu plan with 20 En% fat: A) 7 ± 2 En% linoleic acid (n = 37)
  Interventions: Dietary Supplement: linseed oil
- Linseed oil plus defined background diet (low linolec acid) (Active Comparator): Linseed oil (LO) plus daily menu plans (total dietary fat intake: 30 En%): 10 En% LO plus menu plan with 20 En% fat: B) < 2.5 En% linoleic acid (n = 37)
  Interventions: Dietary Supplement: linseed oil
- Linseed oil plus defined background diet (high milk) (Active Comparator): Linseed oil (LO) plus daily menu plans (total dietary fat intake: 30 En%): 10 En% LO plus menu plan with 20 En% fat: C) 15 ± 2 En% milk fat (n = 37)
  Interventions: Dietary Supplement: linseed oil
- Linseed oil without defined background diet (Placebo Comparator): Linseed oil (LO) without defined menu plans (D) Western diet, n = 37)
  Interventions: Dietary Supplement: linseed oil

INTERVENTIONS:
Dietary Supplement: linseed oil — linseed oil and defined background diet

SUMMARY:
KoALA study - assessment of the influence of the background diet on the metabolism and the bioavailability of plant n-3 PUFA from linseed oil.

In particular, the study design focusses on the impact of variations in the background diet as confounding factor (e.g. variations in concurrently intake of linoleic acid (n-6)). Further, the influence of a regular intake of milk fat, in particular from free-grazing ruminants, on n-3 PUFA metabolism will be investigated.

DETAILED DESCRIPTION:
The KoALA study focuses on the impact of variations in the background diet as a confounding factor. The intake of linoleic acid (LA, C18:2 n-6) has been suggested to diminish the metabolism of α-linolenic acid (ALA, C18:3 n-3) to eicosapentaenoic acid (EPA, C20:5 n-3) and docosahexaenoic acid (DHA, 22:6 n-3).

In this context, the proposed study will be conducted to evaluate the influence of the background diet, in particular the impact of the simultaneous intake of LA on the conversion of ALA into their long-chain (LC) metabolites, the incorporation of n-3 LC-PUFA in human tissues and their metabolism into eicosanoids and docosanoids. Further, the influence of a regular intake of milk fat, in particular from free-grazing ruminants, on n-3 PUFA metabolism will be investigated, because short- and middle-chain fatty acids as well as the branched-chain fatty acids in milk fat may influence the conversion of ALA into n-3 LC-PUFA (hypothesis).

Thus, validated nutrition concepts for increasing n-3 LC-PUFA status from plant sources will be developed to ensure an adequate intake of n-3 PUFA according to the guidelines of nutritional societies and as a contribution to the prevention of cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

Whether participants meet the inclusion criteria will be evaluated by screening prior the run-in (blood sampling).

* Females (in the menopause) and males (50 % each); age: 40 - 65 years; BMI < 30 kg/m2
* Subjects must be able and willing to give written informed consent, and to comply with study procedures
* Subjects with moderate elevated LDL cholesterol (> 3 mmol/l), without lipid-lowering medication
* Persons who consume a traditional "Western diet" composed of meat, sausage, dairy products, cereals, vegetables, fruits etc.
* Precondition: stable eating habits at least one year before enrollment
* Subjects must have adequate fluency in the German language to complete the questionnaires and understand the daily menu plans
* No antihypertensive medication or stable dose for >3 months prior to start of the study and during the entire study period

Exclusion Criteria:

* Subjects with any acute or chronic disease (tumor, infection, other), gastrointestinal diseases, diabe-tes mellitus (type I and II), chronic renal disease, diseases of the parathyroids, diseases necessitat-ing regular phlebotomies other chronic diseases which could affect the results of the present study
* Use of medication which could affect the results of the present study including systemic glucocorti-coids, lipid-lowering medication
* Hormone replacement therapy
* Use of dietary supplements, incl. multivitamins, fish oil capsules, minerals, and trace elements (three months before and during the entire study period)
* Weight loss or weight gain (> 3 kg) during the last three months before study begin
* Relevant food allergies (e.g. milk, nuts etc.)
* Pregnancy or lactation
* Transfusion of blood in the last three months before blood sample taking

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 50 % male, 50 % female (in the menopause)
Enrollment: 148 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2018-07-22 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of EPA and further n-3 PUFA in plasma and erythrocyte lipids | change from baseline after 4, 8 and 12 weeks
  Percentage of EPA and further n-3 PUFA (ALA, DPA, DHA) in plasma and erythrocyte lipids (available from the gas chromatographic analysis)

SECONDARY OUTCOMES:
Fatty acid distribution in plasma lipids | change from baseline after 4, 8 and 12 weeks
  Fatty acid distribution in plasma lipids (including SFA, MUFA, PUFA, > 90 fatty acids) available from the gas chromatographic analysis)
Fatty acid distribution in erythrocyte lipids | change from baseline after 4, 8 and 12 weeks
  Fatty acid distribution in erythrocyte lipids (including SFA, MUFA, PUFA, > 90 fatty acids) available from the gas chromatographic analysis)
Anthropometric and physiological data | change from baseline after 4, 8 and 12 weeks
  height, weight, blood pressure, bioelectrical impedance, waist circumstances, heart rate variability
Blood lipids | change from baseline after 4, 8 and 12 weeks
  total cholesterol, LDL cholesterol, HDL cholesterol, triacylglycerides
Inflammatory markers | change from baseline after 4, 8 and 12 weeks
  eicosanoids, docosanoids
Diabetes risk markers | change from baseline after 4, 8 and 12 weeks
  Insulin, HbA1c, glucose
Clotting markers | change from baseline after 4, 8 and 12 weeks
  alpha prothrombin time, fibrinogen
Cardiovascular risk factors | change from baseline after 4, 8 and 12 weeks
  homocysteine; high sensitive c-reactive protein
Unbound free fatty acid profiles in plasma | change from baseline after 12 weeks
  Unbound free fatty acid profiles in plasma
Futher biomarkers (cardovascular risk factors) | change from baseline after 12 weeks
  Cotinin (marker for smoking), Cystatin C (marker for kidney function), NT-pro-BNP (marker for cardiac function, volume regulation), Troponin (TnT or TnI, marker for myocardial necrosis), Galektin 3 (marker for fibrosis), Asymmetric dimethylarginine (ADMA), homoarginine, trimethylamine N-oxide (TMAO)

CONTACTS AND LOCATIONS:
Locations (1):
- Friedrich-Schiller-University, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: Undecided
publication of the study data and results in national and international journals